CLINICAL TRIAL: NCT07031505
Title: Effects of Photobiomodulation With Superpulsed Laser and Dual Wavelength (810 + 980 NM) in Children and Adolescents With Facial Muscle Pain and Headache: Protocol for a Randomized Controlled Clinical Trial
Brief Title: Effects of Photobiomodulation With Superpulsed Laser and Dual Wavelengths in Children and Adolescents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SuperpulsedLaser
Record Dates: First submitted 2025-06-04; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Facial Pain; Headache
MeSH Terms: conditions — Facial Pain; Headache

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Local photobiomodulation (Experimental): Participants in this arm will receive local photobiomodulation using a high-power superpulsed diode laser (GeminiEvo, Ultradent, USA) with dual wavelengths (810 nm and 980 nm). The protocol consists of 8 sessions (twice weekly for 4 weeks), with laser applied to the masseter, temporal, trapezius, and temporomandibular joint (TMJ) regions. Each point will be irradiated for 13 seconds using 4 J of energy (10.52 J/cm²) with a contact technique. Safety procedures include use of protective eyewear and disinfection of the device tip.
  Interventions: Device: Active Photobiomodulation
- Group 2 - Sham local photobiomodulation (Sham Comparator): Participants in this arm will undergo the same treatment protocol as the experimental group. However, the device will be deactivated (no laser emission), while maintaining the guide light and operational sounds to ensure participant blinding. All application parameters and session conditions will mimic the active group.
  Interventions: Device: Sham Photobiomodulation

INTERVENTIONS:
Device: Active Photobiomodulation — Local photobiomodulation using a high-power superpulsed diode laser (GeminiEvo, Ultradent, USA) with dual infrared wavelengths (810 nm and 980 nm). Eight sessions will be conducted (twice a week for 4 weeks). Application will be at one point each on the masseter, temporal, trapezius, and temporomandibular joint regions. Each point will be irradiated for 13 seconds with 4 J of energy (10.52 J/cm²), in contact mode. The procedure includes safety measures such as protective eyewear and disinfection of the laser tip.
  Arms: Group 1 - Local photobiomodulation
Device: Sham Photobiomodulation — The same application protocol as the experimental group will be followed, using the same laser device (GeminiEvo, Ultradent, USA), but with the laser emission deactivated. The guide light and sound will remain active to preserve participant blinding. Application points, duration, frequency, and session environment will be identical to the active group.
  Arms: Group 2 - Sham local photobiomodulation

SUMMARY:
This randomized clinical trial evaluates the effects of photobiomodulation with a superpulsed diode laser (810 + 980 nm) on orofacial pain and tension-type headache in children and adolescents. Sixty participants will be assigned to receive active PBM or sham therapy over eight sessions. Pain and anthropometric variables will be assessed.

DETAILED DESCRIPTION:
Orofacial pain and tension-type headache are common in children and adolescents, often impairing school performance, social interactions, and functional development. Due to potential side effects of pharmacological treatments, non-pharmacological alternatives like photobiomodulation (PBM) are being studied. This protocol evaluates the effects of PBM with a superpulsed dual-wavelength diode laser (810 nm + 980 nm) applied to masseter and temporal muscles across eight sessions. Sixty participants (aged 6-17) will be randomized into two groups: G1 (active PBM) and G2 (sham). Anthropometric data (age, weight, height, BMI, Fitzpatrick phototype), penetrated energy, and local temperature will be recorded. Pain will be assessed using the Faces Pain Scale and the ICHD-3 questionnaire. The primary outcome is pain reduction. Secondary outcomes include correlations between anthropometric factors, energy penetration, and clinical response. A linear mixed model with repeated measures will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents 6 to 17 years of age enrolled at the medical and dental clinic of Universidade Nove de Julho (UNINOVE), Vergueiro Campus;
* Children and adolescents who present with at least one symptom of orofacial pain and/or headache, according to the Faces Pain Scale and the childhood and adolescence headache questionnaire based on the ICHD-3

Exclusion Criteria:

* Pregnant adolescents;
* Having taken corticoids, non-steroidal anti-inflammatory drugs or analgesics in the previous 30 days;
* Having taken isotretinoin;
* Individuals who report photosensitivity to laser or LED in previous treatments.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity based on Faces Pain Scale | Weekly, up to 4 weeks
  The Faces Pain Scale will be completed weekly by the legal guardians during the second therapeutic session of each treatment week.
Headache classification using ICHD-3 | Weekly, up to 4 weeks
  The ICHD-3 questionnaire will be completed weekly by the legal guardians during the second therapeutic session of each treatment week.

SECONDARY OUTCOMES:
Light transmission | Day 1
  Light transmission will be assessed through each participant's index finger and cheek (masseter muscle) using a SPER Scientific Pocket Laser Power Meter. The measurement will follow the Yaroslavsky method and will be collected during the first treatment session.
Local temperature | Day 1
  Temperature will be measured using a dual infrared laser thermometer during the first treatment session, specifically during the application of photobiomodulation.